CLINICAL TRIAL: NCT04084106
Title: Effects of Phenoximethylpenicillin, Amoxicillin and Amoxicillin-clavulanic Acid on the Gut Microbiota of Healthy Volunteers: a Randomized Clinical Trail
Brief Title: Effects of Phenoximethylpenicillin, Amoxicillin and Amoxicillin-clavulanic Acid on the Gut Microbiota
Acronym: EPAAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Thomas Tängdén, Associate professor, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-03300
Record Dates: First submitted 2019-08-30; First posted 2019-09-10 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Infectious Disease
Keywords: randomized trial; antibiotic resistant genes; gut microbiota; healthy volunteers; metagenomics
MeSH Terms: conditions — Communicable Diseases | interventions — Penicillin V; Amoxicillin; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Intervention Model Description: Randomized clinical trail
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- phenoximethylpenicillin (Experimental): phenoximethylpenicillin, tablet, 1 g 3 times daily for 5 days.
  Interventions: Drug: Phenoxymethylpenicillin
- amoxicillin (Active Comparator): amoxicillin, tablet, 500 mg 3 times daily for 5 days.
  Interventions: Drug: Amoxicillin
- amoxicillin-clavulanic acid (Active Comparator): amoxicillin-clavulanic acid tablet, 500/125 mg 3 times daily for 5 days.
  Interventions: Drug: Amoxicillin-clavulanic acid
- No intervention (No Intervention): No intervention

INTERVENTIONS:
Drug: Phenoxymethylpenicillin — Oral administration
  Arms: phenoximethylpenicillin
Drug: Amoxicillin — Oral administration
  Arms: amoxicillin
Drug: Amoxicillin-clavulanic acid — Oral administration
  Arms: amoxicillin-clavulanic acid

SUMMARY:
The overall aim of the project is to fill an important knowledge gap on the ecological effects of selected antibiotics. The results will be used to guide treatment decisions for common infections to as much as possible reduce the negative impact on the intestinal microbiota and consequently the risks of side effect and resistance development during therapy.

Specific aims for this study are to determine (1) the composition of intestinal microbiota and prevalence of resistant bacteria and resistance genes prior to and up to 1 year after antibiotic treatment, and (2) the relative effects on the microbiota after treatment with three antibiotics used for lower respiratory tract infections; phenoximethylpenicillin, amoxicillin and amoxicillin-clavulanic acid, or no treatment (control).

A total of 120 healthy volunteers will be recruited to the study. They are randomised to 5 days' treatment with phenoximethylpenicillin, amoxicillin or amoxicillin-clavulanic acid, or to no antibiotic treatment. Subjects submit faecal samples at eight different time-points; at the start of the study (before treatment), immediately, one week and 1, 3, 6, 12 and 24 months after completion of the treatment. The samples will be delivered to Scilifelab for metagenomic sequencing to detect antibiotic resistant genes and analysis of the intestinal microbiota and to the Microbiology ward for analysis with phenotypic methods (culturomics) to detect resistant genes and resistant bacteria.

DETAILED DESCRIPTION:
Background: The rationale behind this project is that different antibiotics have varying effects on the intestinal microbiota, which has clinical implications. To investigate the relative collateral damage during treatment with different antibiotics a randomized trial is needed. Repeated sampling during a 1-year period is required to capture prolonged disturbance and the time to a restored microbiota. To readily examine the antibiotic effects healthy volunteers are ideal for the study as their microbiota is most likely to be normal at inclusion. They also have a low risk of encountering other factors during follow-up that will affect the composition of the intestinal bacteria.

Aim: The purpose of the study is to determine: (1) composition of intestinal microbiota and prevalence of resistant bacteria and resistance genes prior to and up to 1 year after antibiotic treatment, and (2) differences in the microbiota after treatment with antibiotics; phenoximethylpenicillin, amoxicillin and amoxicillin-clavulanic acid respectively compared to no treatment.

Method: The study is a conducted within the Department of Infectious Diseases at Uppsala University Hospital. A total of 120 healthy volunteers will be recruited to the study. They are randomised to 5 days' treatment with phenoximethylpenicillin, amoxicillin or amoxicillin-clavulanic acid, or to no antibiotic treatment. Subjects submit faecal samples at eight different time-points; at the start of the study (before treatment), immediately, one week and 1, 3, 6, 12 and 24 months after completion of the treatment. Altogether, the subjects will provide 8 faecal samples during the course of the study. A total of 960 faecal samples will be collected and analysed.

Each subject will submit two faecal samples at each time-point. One sample will be frozen in DNA-shield and delivered to Scilifelab for analysis of the intestinal microbiota and metagenomic sequencing to detect antibiotic resistant genes.The other faecal sample will be delivered to the Microbiology department for analysis with phenotypic methods (culturomics) to detect resistant genes and resistant bacteria.

Statistics: The compilation of data and statistics will primarily be descriptive. We will analyse the intestinal microbiota and the prevalence of resistance genes in the subjects prior to and immediately after antibiotic treatment, and then monitor the composition (diversity) of the intestinal microbiota, resistant bacteria and resistance genes 1 week, 1, 3, 6, 12 and 24 months after completion of the treatment. Diversity will be analysed using metagenomics (shotgun) and is used as a variable to compare the degree of collateral damage on the intestinal microbiota with different antibiotics, and to compare the intestinal microbiota before and after antibiotic treatment in the same individual. The diversity of the intestinal microbiota in faecal sample 1 will constitute the baseline. Targeted statistical calculations on differences between treatment groups and gender as regards intestinal microbiota, resistance and side effects will be carried out depending on outcomes, which cannot be predicted in advance.

Endpoints and outcomes: The primary endpoint is the diversity and composition of the intestinal microbiota, the prevalence of multidrug-resistant Gram-negative bacteria in screening cultures and the prevalence of antibiotic resistance genes in faeces prior to and up to 2 year after antibiotic treatment.

The results may be used as a basis for targeting the choice of antibiotic for pulmonary infections (pneumonia) towards those antibiotics that have the least risk of disrupting the intestinal microbiota and leading to resistance.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Age ≥ 18 years

Exclusion Criteria:

* Chronic disease, allergy, asthma, recurrent infections
* Ongoing antibiotic treatment
* Antibiotic treatment the past 12 months
* Pregnancy or planned pregnancy within the study period
* Known allergy to phenoximethylpenicillin, amoxicillin and amoxicillin- clavulanic acid
* Planned travel outside Europe within one year from inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Diversity of the intestinal microbiota prior to and after (any) antibiotic treatment as determined with metagenomics on repeated faecal samples. | 2 year
  The diversity of the intestinal microbiota prior to and up to 2 year after antibiotic treatment will be determined by sequencing with shotgun metagenomics.
Comparison of the diversity of the intestinal microbiota with three different antibiotics - phenoxymethylpenicillin (reference), amoxicillin and amoxicillin-clavulanic acid - as determined with metagenomics on repeated faecal samples. | 2 years
  The relative effects of on the diversity of the intestinal microbiota prior to and up to 2 year after antibiotic treatment will be determined by sequencing with shotgun metagenomics.
Prevalence of resistance genes in the intestinal microbiota prior to and after (any) antibiotic treatment as determined with metagenomics on repeated faecal samples. | 2 years
  The prevalence of resistant bacteria and resistance genes prior to and up to 2 year after antibiotic treatment will be determined by sequencing with shotgun metagenomics.
Comparison of the prevalence of resistance genes in the intestinal microbiota with different antibiotics - phenoxymethylpenicillin, amoxicillin and amoxicillin-clavulanic acid - as determined with metagenomics on repeated faecal samples. | 2 years
  The relative effects of on the prevalence of resistant bacteria and resistance genes prior to and up to 2 year after treatment with phenoxymethylpenicillin (reference), amoxicillin or amoxicillin-clavulanic acid will be determined by sequencing with shotgun metagenomics.
Prevalence of multidrug-resistant bacteria in the intestinal microbiota prior to and after (any) antibiotic treatment as determined with phenotypic analyses on repeated faecal samples. | 2 years
  Multidrug-resistant gram-negative bacteria will be isolated and characterized by incubation in selective media, MIC determination using conventional methods and PCR/whole-genome sequencing to determine the presence of resistance genes.
Comparison of the prevalence of resistant bacteria in the intestinal microbiota with three different antibiotics - phenoxymethylpenicillin, amoxicillin and amoxicillin-clavulanic acid - as determined with phenotypic analyses on repeated faecal samples. | 2 years
  Multidrug-resistant gram-negative bacteria producing will be isolated and characterized by incubation in selective media, MIC determination using conventional methods and PCR/whole-genome sequencing to determine the presence of resistance genes.

SECONDARY OUTCOMES:
Prevalence of adverse events with (any) antibiotic treatment. | 1 year
  Information on side effects during and following antibiotic treatment will be collected using diaries and questionnaires.
Comparison of prevalence of adverse events with three different antibiotics - phenoxymethylpenicillin (reference), amoxicillin and amoxicillin-clavulanic acid. | 1 year
  Information on side effects during and following antibiotic treatment will be collected using diaries and questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Tängdén, MD, PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden